CLINICAL TRIAL: NCT02104401
Title: Pilot Study: Open Label Treatment With tDCS for Parkinson's and Related Disorders for Improvement of Speech, Gait and Mood
Brief Title: Open Label Treatment With tDCS for Parkinson's and Related Disorders for Improvement of Speech, Gait and Mood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Ferrell Family Charitable Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00000
Record Dates: First submitted 2014-04-02; First posted 2014-04-04 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tDCS (Experimental): tDCS will be applied with a Soterix CT tDCS Device with a HD-tDCS 4x1 Multi-Channel Stimulation Interface. During stimulation, a low level of constant DC electrical current (1-2 mA) will be applied via the electrodes. Current will be ramped up over 10-60 seconds, and typically causes very mild tingling and itching sensations. The current will be applied for no more than 20 minutes per session, at which time the current is ramped down over 10-60 seconds. Subjects will be seated in a chair throughout tDCS administration. Subjects will receive tDCS 5 days/week for 4 weeks.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — tDCS will be applied with a Soterix CT tDCS Device with a HD-tDCS 4x1 Multi-Channel Stimulation Interface. During stimulation, a low level of constant DC electrical current (1-2 mA) will be applied via the electrodes. Current will be ramped up over 10-60 seconds, and typically causes very mild tingling and itching sensations. The current will be applied for no more than 20 minutes per session, at which time the current is ramped down over 10-60 seconds. Subjects will be seated in a chair throughout tDCS administration. Subjects will receive tDCS 5 days/week for 4 weeks.

SUMMARY:
This research will help us to understand whether transcranial direct current stimulation (tDCS) can safely improve recovery of speech and language abilities, gait , and mood in people with Parkinson's disease and related disorders. Some of the disorders that will be studied to understand if tDCS can be useful include Parkinson's Disease, Multi-System Atrophy (MSA) and progressive supranuclear palsy (PSP).

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease or a related disorder (e.g. Multiple Systems Atrophy) as diagnosed by a neurologist specializing in Movement Disorders
* Age >= 18 years

Exclusion Criteria:

* Skull defect at or near site of tDCS delivery.
* History of a significant stroke or traumatic brain injury.
* History of other brain conditions that could impact interpretation of results (such as MS, brain tumor, encephalitis).
* Presence of implanted electrical or metallic devices in the head or body (examples include cardiac pacemakers or defibrillators, Baclofen pumps, deep brain stimulators, ventricular shunts with metallic parts, vagus nerve stimulators)
* Presence of ferrous metal in the head (except titanium; for instance shrapnel)
* History of psychiatric disease requiring hospitalization, electroconvulsive therapy, or ongoing medication use (other than common antidepressants)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Improvement of Motor and Speech Symptoms of Parkinson's Disease or Related Disorders | 16 weeks
  We will perform an assessment of motor function using Part III of the Unified Parkinson's Disease Rating Scale (UPDRS), timed test of gait, and patient self-assessment. Speech functions will be assessed with sentence repetition,evaluation of spontaneous speech, and other standard language tests. The assessment will also include other measures and questionnaires (e.g. Bech Depression Inventory) to be filled out by the patient and his/her family.

SECONDARY OUTCOMES:
Improvement of Neuropsychiatric Symptoms of Parkinson's Disease or Related Disorders | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Pagan, MD, Principal Investigator — Georgetown University
Locations (1):
- MedStar Georgetown University Hospital, Washington D.C., District of Columbia, United States